CLINICAL TRIAL: NCT00077012
Title: A Phase I/II Dose Escalation Study to Assess the Safety, Tolerability, and Preliminary Efficacy of Transurethral Photodynamic Therapy With QLT0074 for Benign Prostatic Hyperplasia
Brief Title: Dose Escalation Study With QLT0074 for Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPH 002
Record Dates: First submitted 2004-02-09; First posted 2004-02-11 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — QLT0074; Photochemotherapy

INTERVENTIONS:
Drug: QLT0074
Drug: Photodynamic therapy

SUMMARY:
The primary objective of this study is to assess the safety and tolerance of transurethral photodynamic therapy (PDT) with QLT0074.

Secondary objectives are:

1. To determine if transurethral PDT with QLT0074 has a therapeutic effect on benign prostatic hyperplasia (BPH), evaluated by the American Urological Association Symptom Index (AUA SI), urinary flow rate (Qmax), and post-void residual volume (PVR).
2. To determine the extent of systemic exposure to QLT0074 following transurethral intraprostatic injection.
3. To select up to two transurethral PDT drug-light regimens for further clinical development.

DETAILED DESCRIPTION:
This will be a multicenter, uncontrolled, dose escalation, exploratory study in subjects with symptomatic BPH. Six study centers are planned.

Each subject will receive a fixed dose of QLT0074 (0.4 mg) injected transurethrally into the prostate followed by transurethral light application to activate the drug. Five light dose cohorts will be investigated sequentially (25, 50, 80, 120, and 150 J/cm2), with 3 subjects in the first cohort and 6 subjects in cohorts 2-5 for a total of 27 subjects. The follow-up period for each subject is 180 days. There will be a minimum 30-day interval between treatment of the last subject in one cohort (Day 0) and treatment of the first subject in the next cohort to monitor predefined toxicities and ensure safety and tolerance in subjects of the previous cohort.

A Safety Monitoring Committee will evaluate toxicity related to PDT effects, and approve escalation of the light dose for each cohort. The light dose will not be escalated if any of the following predefined toxicity criteria occur and are judged to be related to a PDT effect by the Safety Monitoring Committee:

1. 1 or more subjects in the cohort experience macroscopic urinary bleeding not resolved by Day 14, or
2. 2 or more subjects in the cohort experience intolerable urinary pain not controlled with over-the-counter medication by Day 14, or
3. 1 or more subjects in the cohort experience any other clinically significant urological adverse event, as judged by the Investigator and confirmed by the Safety Monitoring Committee.

In addition to the above events, the Safety Monitoring Committee will evaluate the incidence, timing, severity, and frequency of other adverse events and serious adverse events to assess the safety of transurethral PDT and the treatment procedures (such as the use of the cystoscope, InjectTx device, treatment balloon-catheter, etc).

To prevent treating subjects with a light dose greater than that which already provides substantial clinical benefit, the Safety Monitoring Committee will review preliminary efficacy data (AUA SI scores and Qmax values) after all subjects in a cohort (for each of the first 4 cohorts) have completed the Day 90 visit. Further enrollment will be curtailed if more than 75% of subjects in a cohort experience both of the following efficacy stopping criteria by Day 90:

1. greater or equal to 75% reduction in the AUA SI score and,
2. greater or equal to 100% increase in Qmax.

ELIGIBILITY:
* Twenty-seven men with symptomatic BPH despite adequate drug therapy and who are candidates for surgical or minimally invasive treatment will be enrolled in the study.
* Subjects must have an AUA SI >13, Qmax between 5 and 15 mL/sec, and a urethral treatment length between 30 and 65 mm (defined as the length of the urethra between the bladder neck and the edge of the verumontanum distal to the bladder).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Raymond Fay, MD, Inc, San Francisco, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - North Texas Veteran Affairs Health Care System, Dallas, Texas
- Canada (2):
  - The Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - Royal Victoria Hospital, Montreal, Quebec